CLINICAL TRIAL: NCT03302195
Title: Optimal Cardiopulmonary Bypass and Anticoagulation Management Strategies in Obese Patients Undergoing Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Pierre Voisine, Cardiac surgeon, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obesity-CPB-21117
Record Dates: First submitted 2017-09-28; First posted 2017-10-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Cardiopulmonary Bypass; Obesity
Keywords: Heparin; Allogeneic blood product transfusions; Bleeding; Cardiac surgery; Obesity
MeSH Terms: conditions — Obesity; Hemorrhage | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Randomized control prospective trial
Who Masked: Participant
Masking Description: Participant is blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Active Comparator): Heparin dose and cardiopulmonary bypass pump flow rate are calculated using total body weight.
  An initial 400 IU/Kg Heparin dose will be administered, with an additional dose of 75 IU/kg if the activated clotting time remains below the 425 seconds target value. The cardiopulmonary bypass pump flow rate of 2.4 L/min/m2 of body surface area will be calculated.
  Interventions: Drug: Heparin; Procedure: cardiopulmonary bypass pump flow rate
- Intervention group A (Experimental): Heparin dose is adjusted for lean body weight and cardiopulmonary bypass pump flow rate is calculated using total body weight.
  An initial 400 IU/Kg Heparin dose will be administered, with an additional dose of 75 IU/kg if the activated clotting time remains below the 425 seconds target value. The cardiopulmonary bypass pump flow rate of 2.4 L/min/m2 of body surface area will be calculated.
  Interventions: Drug: Heparin; Procedure: cardiopulmonary bypass pump flow rate
- Intervention group B (Experimental): Heparin dose is calculated using total body weight and cardiopulmonary bypass pump flow rate is adjusted for lean body weight.
  An initial 400 IU/Kg Heparin dose will be administered, with an additional dose of 75 IU/kg if the activated clotting time remains below the 425 seconds target value. The cardiopulmonary bypass pump flow rate of 2.4 L/min/m2 of body surface area will be calculated.
  Interventions: Drug: Heparin; Procedure: cardiopulmonary bypass pump flow rate
- Intervention group C (Experimental): Heparin dose and cardiopulmonary bypass pump flow rate are adjusted for lean body weight.
  An initial 400 IU/Kg Heparin dose will be administered, with an additional dose of 75 IU/kg if the activated clotting time remains below the 425 seconds target value. The cardiopulmonary bypass pump flow rate of 2.4 L/min/m2 of body surface area will be calculated.
  Interventions: Drug: Heparin; Procedure: cardiopulmonary bypass pump flow rate

INTERVENTIONS:
Drug: Heparin — Based on patient body weight (UI/kg)
Procedure: cardiopulmonary bypass pump flow rate — Based on patient body weight (L/min/m2)

SUMMARY:
Standard Heparin management, based on total body weight, is not well established for obese patients undergoing cardiac surgery with cardiopulmonary bypass (CPB).

The purpose of this study is to assess the safety and efficacy of using lean body mass (LBM) to determine pump flow rate and/or Heparin dosage in obese patients undergoing CPB.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI ≥ 30kg/m2)
* Planned cardiac surgery
* Age ≥ 18 years

Exclusion Criteria:

* Permanent pacemaker
* Known intolerance to protamine
* Known or suspected allergy to the used antifibrinolytic agent
* Refusal to receive blood products
* Planned off pump coronary artery bypass
* Planned peri-operative use of desmopressin
* Known Heparin-induced thrombocytopenia
* Known deficiency in protein C, protein S, antithrombin or homozygous factor V Leiden
* Known congenital bleeding disorders
* Current endocarditis
* Planned hypothermic circulatory arrest (<28C)
* Two or more cardiac surgery procedures
* Emergency cardiac surgery procedures (medically required within 24hours of presenting with acute symptoms)
* Planned CPB priming with red blood cells
* Any known autoimmune disease
* Any history of stroke or non-coronary thrombotic disorders including deep venous thrombosis and pulmonary embolism
* Significant (≥50%) carotid artery stenosis
* Patient dosed with low molecular weight Heparin less than 24h before surgery
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Confirmed ST elevation myocardial infarction (STEMI) within 7 days
* Pre-operative platelet count <100,000/microliter
* Anaemia (Hematocrit <32% for females, <35%for males)
* Dosed with clopidogrel or ticagrelor within the last 5 days prior to surgery, or prasugrel within 7 days
* Dosed with GPIIb/IIIa receptor blockers (Abciximab, Tirofiban, Eptifibatide) ≤ 24 hours prior to surgery
* International ratio (INR) >1.5 on the day of surgery in patients treated with vitamin K antagonist
* Liver dysfunction (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) increased ≥ 2-fold above the upper limit of local laboratory normal ranges)
* Renal failure (creatinine ≥ 175 micromol/L or dialysis)
* Current thromboembolic disease other than myocardial infarct
* Patients who have pre-donated autologous blood
* Patient presenting with a resistance to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2015-08-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Allogeneic transfusions of red blood cells | Seven days post-operatively or until discharge, whichever comes first
  Percentage of subjects avoiding any allogeneic transfusions of red blood cells

SECONDARY OUTCOMES:
Allogeneic transfusions of blood products | Seven days post-operatively or until discharge, whichever comes first
  Percentage of subjects avoiding any allogeneic transfusions
Units of blood product transfusions | Seven days post-operatively or until discharge, whichever comes first
  Number of units of transfused blood products
Massive red blood cell transfusions | Seven days post-operatively or until discharge, whichever comes first
  Percentage of subjects avoiding massive red blood cell transfusion (more than 5 units)
Post-operative complications | Post-operatively from day 0 up to first hospital discharge
  Monitoring the safety of strategies by monitoring post-operative complications
Bleeding | Peroperative, 4 and 24 hours post-operative
  Per- and post-operative bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Voisine, MD, Principal Investigator — University Laval
Locations (1):
- Hopital Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No